CLINICAL TRIAL: NCT00660491
Title: Endothelial Dysfunction Induced by Postprandial Lipemia: Complete Protection Afforded by High Intensity Aerobic Interval Exercise
Brief Title: Endothelial Dysfunction Induced by Postprandial Lipemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Exercise, Food and Endothelium
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Healthy Subjects
Keywords: flow mediated dilatation; maximal oxygen uptake; blood lipid
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): Control
- 2 (No Intervention): moderate exercise training group
- 3 (Experimental): high intensity exercise group
  Interventions: Other: exercise training

INTERVENTIONS:
Other: exercise training — moderate intensity exercise group, and high intensity exercise group
  Arms: 3

SUMMARY:
Postprandial lipemia and exercise oppose each other in terms of cardiovascular risk, however the mechanism of their interaction is not well understood.

Therefore we want to study vascular function, as assessed by brachial artery (BA) flow mediated dilation (FMD), in healthy men before and after a high fat meal (HFM) preceded (16-18 hrs) by rest, a single bout of continuous moderate intensity exercise (CME), and high intensity interval exercise (HIIE).

ELIGIBILITY:
Inclusion Criteria:

* male, 20-40years, BMI between 25 and 30, resident in Trondheim.

Exclusion Criteria:

* unstable angina, CHD, heart failure,

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilatation | baseline, post exercise, 30min, 2hour, 4hour post exercise

SECONDARY OUTCOMES:
blood lipid profile | same as flow mediated dilatation

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisloff, Professor, Study Chair — National Taiwan Normal University
Locations (1):
- NTNU, Trondheim, Norway

REFERENCES:
- [Result] Tyldum GA, Schjerve IE, Tjonna AE, Kirkeby-Garstad I, Stolen TO, Richardson RS, Wisloff U. Endothelial dysfunction induced by post-prandial lipemia: complete protection afforded by high-intensity aerobic interval exercise. J Am Coll Cardiol. 2009 Jan 13;53(2):200-6. doi: 10.1016/j.jacc.2008.09.033. PMID 19130989